CLINICAL TRIAL: NCT04732494
Title: A Phase 2, Multicenter, Randomized, Placebo-Controlled Study to Compare the Efficacy of Anti-PD-1 Monoclonal Antibody Tislelizumab (BGB-A317) Plus Anti-TIGIT Monoclonal Antibody Ociperlimab (BGB-A1217) Versus Tislelizumab Plus Placebo as Second-Line Treatment in Patients With PD-L1 Tumor Area Positivity (TAP) ≥ 10% Unresectable, Locally Advanced, Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Brief Title: Anti-PD-1 Monoclonal Antibody Tislelizumab (BGB-A317) Combined With or Without Anti-TIGIT Monoclonal Antibody Ociperlimab (BGB-A1217) in Participants With Recurrent or Metastatic Esophageal Squamous Cell Carcinoma
Acronym: AdvanTIG-203
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BGB-A317-A1217-203; 2020-004658-32 (EudraCT Number); CTR20213241/CTR20210243 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-01-25; First posted 2021-02-01 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2024-12

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — tislelizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Tislelizumab plus Ociperlimab (Experimental): Participants received 200 milligrams (mg) tislelizumab plus 900 mg ociperlimab intravenously once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
  Interventions: Biological: Tislelizumab; Biological: Ociperlimab
- Arm B: Tislelizumab plus Placebo (Placebo Comparator): Participants received 200 mg tislelizumab plus placebo intravenously once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
  Interventions: Biological: Tislelizumab; Drug: Placebo

INTERVENTIONS:
Biological: Tislelizumab — Tislelizumab is a monoclonal antibody formulated for intravenous injection.
  Other Names: BGB-A317; TEVIMBRA®
Biological: Ociperlimab — Ociperlimab is a monoclonal antibody formulated for intravenous injection.
  Other Names: BGB-A1217
  Arms: Arm A: Tislelizumab plus Ociperlimab
Drug: Placebo — Ociperlimab placebo injection is a sterile, preservative-free solution for infusion formulated in the same buffer as ociperlimab active drug.
  Other Names: Ociperlimab placebo
  Arms: Arm B: Tislelizumab plus Placebo

SUMMARY:
A study of tislelizumab (BGB-A317) plus ociperlimab versus tislelizumab plus placebo as second-line treatment in participants with programmed cell death protein-ligand 1 (PD-L1) tumor area positivity (TAP) ≥ 10% unresectable, locally advanced, recurrent or metastatic esophageal squamous cell carcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed diagnosis of esophageal squamous cell carcinoma (ESCC).
2. Have progressive disease during or after first-line of systemic treatment for unresectable, locally advanced, recurrent or metastatic ESCC.
3. Have measurable disease as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
4. Have confirmed programmed cell death protein-ligand 1 (PD-L1) tumor area positivity (TAP) ≥ 10% in tumor tissues tested by the central lab.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.

Key Exclusion Criteria:

1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, T-cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine-based inhibitory motif domains, or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways.
2. Participants with evidence of fistula (either esophageal/bronchial or esophageal/aorta).
3. Evidence of complete esophageal obstruction not amenable to treatment.
4. Uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage (recurrence within 2 weeks after intervention).
5. Has received any chemotherapy, immunotherapy (eg, interleukin, interferon, thymosin, etc) or any investigational therapies within 14 days or 5 half-lives (whichever is longer) before the first dose of study drug. Or has received palliative radiation treatment or other local regional therapies within 14 days before the first dose of study drug.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (86):
- China (52):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Quanzhou First Hospital of Fujian Province, Quanzhou, Fujian
  - First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Lanzhou University Second Hospital, Gansu, Gansu
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Meizhou Hospital Affiliated to Sun Yat-sen University, Guangzhou, Guangdong
  - Hainan Third People's Hospital, Sanya, Hainan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai Provincial People's Hospital, Qinghai, Qinghai
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - People's Hospital of Deyang City, Deyang, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - First Affiliated Hospital of Kunming Medical University, Yunnan, Yunnan
  - Beijing Cancer Hospital, Beijing
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - The First People's Hospital of Changzhou, Changzhou
  - Fujian Cancer Hospital, Fujian
  - The First Affiliated Hospital of Fujian Medical University, Fujian
  - Zhongshan Hospital Xiamen University, Fujian
  - Cancer Hospital of Shantou University Medical College, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangdong
  - Sun Yat-sen University Cancer Center, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangdong
  - The Sixth Affiliated Hospital, Sun Yat-sen University, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Guangxi
  - Hainan General Hospital, Hainan
  - Affiliated Hospital of Hebei University, Hebei
  - The Second Hospital of Anhui Medical University, Hefei
  - Harbin Medical University Cancer Hospital, Heilongjiang
  - Henan Cancer Hospital, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Henan
  - The First Affiliated Hospital of Zhengzhou University, Henan
  - Hubei Cancer Hospital, Hubei
  - Xiangyang Central Hospital, Hubei
  - Hunan Cancer Hospital, Hunan
  - The First Affiliated Hospital of Nanchang University, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Jiangxi
  - Linyi Cancer Hospital, Shandong
  - Weifang People's Hospital, Shandong
  - Shanghai Chest Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Sichuan Provincial People's Hospital, Sichuan
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Hangzhou Cancer Hospital, Zhejiang
  - Hwa Mei Hospital, University of Chinese Academy of Sciences, Zhejiang
- France (4):
  - Centre Hospitalier Universitaire d'Amiens - Hopital Sud, Amiens, Picardie
  - Hôpital de la Timone, Marseille
  - Hopital Europeen Georges Pompidou - Digestive Oncology, Paris
  - CHU de Poitiers, Poitiers
- South Korea (8):
  - Ajou University Hospital, Gyeonggi-do
  - Chonnam National University Hwasun Hospital, Jeongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Institut Catala D'Oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Clinico Universitario de Valencia - Incliva, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (6):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (6):
  - Chulabhorn Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai University, Chiang Mai
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 52 study centers in 7 countries/regions in Chinese mainland, Chinese Taiwan, South Korea, Thailand, France, Spain, and Russia.
Pre-assignment Details: Participants were randomized equally to one of two treatment groups. Randomization was stratified by Eastern Cooperative Oncology Group Performance Status (ECOG PS) score (0 versus 1), number of organs with metastases (≤ 1 versus ≥ 2), and region (Asia versus non-Asia).
Period: Overall Study
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Started | 62 | 63
Received Treatment Plan | 62 | 63
Completed | 0 | 0
Not Completed | 62 | 63
Not completed — Death | 39 | 36
Not completed — Study Closed by Sponsor | 20 | 15
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Lost to Follow-up | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Arm A: Tislelizumab Plus Ociperlimab: Participants received 200 mg tislelizumab plus 900 mg ociperlimab intravenously once every 3 weeks until disease progression, unacceptable toxicity, or withdrawal of informed consent, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 27 | 67
  >=65 years | 22 | 36 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (7.31) | 63.6 (7.33) | 62.5 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 58 | 53 | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 56 | 54 | 110
  White | 3 | 5 | 8
  Not Reported | 3 | 3 | 6
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG Performance Status is used to assess a patient's disease status, and how the disease affects daily living activities according to the following scale:
  0 = Fully active, able to carry out all activities without restriction;
  1. = Restricted in physically strenuous activity, ambulatory and able to carry out work of a light nature;
  2. = Ambulatory and capable of all self-care, unable to carry out any work activities. Up and about > 50% of waking hours;
  3. = Capable of only limited self-care, confined to bed or chair > 50% of waking hours;
  4. = Completely disabled, confined to bed or chair.
  Participants
    0 (Fully active) | 16 | 15 | 31
    1 (Restricted but ambulatory) | 46 | 48 | 94
Number of Organs With Metastases [Count of Participants; unit: Participants]
  ≤ 1 organ | 32 | 33 | 65
  ≥ 2 organs | 30 | 30 | 60
Region [Count of Participants; unit: Participants]
  Asia | 54 | 54 | 108
  Non-Asia | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Assessed by the Investigator
Description: Objective response rate is defined as the percentage of participants who had a best overall response of confirmed complete response (CR) or partial response (PR) assessed by the Investigator according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
  Response evaluations were performed using computed tomography or magnetic resonance imaging (MRI) approximately every 6 weeks for the first 54 weeks and then every 12 weeks thereafter.
  CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) < 10 mm, and no new lesions.
  PR: At least a 30% decrease in the size of target lesions, with no progression of non-target lesions and no new lesions, or disappearance of target lesions with persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions.
  Response (CR or PR) must have been confirmed 4 weeks or later after the first response was observed.
Time Frame: Up to the primary analysis data cutoff date of 01 February 2023; median (range) time on follow-up was 7.4 (0.5 - 20.1) months in Arm A and 6.4 (0.4 - 20.2) months in Arm B.
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
percentage of participants | 30.6 [19.6 to 43.7] | 20.6 [11.5 to 32.7]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Test type: Superiority — The primary endpoint ORR was tested at a 2-sided alpha of 0.05; p = 0.2114, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel method stratified by the stratification factors (ECOG PS score [0 vs 1] and number of organs with metastases [≤ 1 vs ≥ 2]); Risk Difference (RD) = 9.9, 95% CI 2-sided [-5.4 to 25.3] — Mantel-Haenszel common risk difference stratified by the stratification factors (ECOG PS score [0 vs 1] and number of organs with metastases [≤ 1 vs ≥ 2])

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) is defined as the time from the date of randomization until the date of death due to any cause.
  Median overall survival was estimated using the Kaplan-Meier method. For participants who were still alive at the end of the trial, OS was censored at the last known alive date or the date of data cutoff, whichever was earlier.
Time Frame: From randomization to the end of the study, median (range) time on follow-up was 10.0 (0.5 - 29.9) months in Arm A and 7.8 (0.4 - 29.3) months in Arm B.
Population: The Intent-to-Treat Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
months | 10.2 [7.9 to 19.5] | 9.3 [6.4 to 14.8]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Test type: Other; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.58 to 1.45] — Hazard ratio and 95% confidence intervals (CIs) were estimated using a Cox regression model stratified by the selected stratification factors (ECOG PS score [0 vs 1] and the number of organs with metastases [≤ 1 vs ≥ 2])

3. Secondary Outcome: Objective Response Rate Assessed by the Independent Review Committee
Description: Objective response rate is defined as the percentage of participants who had a best overall response of confirmed complete response (CR) or partial response (PR) assessed by the Independent Review Committee (IRC) according to RECIST v1.1.
  Response evaluations were performed using computed tomography or MRI approximately every 6 weeks for the first 54 weeks and then every 12 weeks thereafter.
  CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) < 10 mm, and no new lesions.
  PR: At least a 30% decrease in the size of target lesions, with no progression of non-target lesions and no new lesions, or disappearance of target lesions with persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions.
  Response (CR or PR) must have been confirmed 4 weeks or later after the first response was observed.
Time Frame: as for outcome 1
Population: The Intent-to-Treat Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
percentage of participants | 32.3 [20.9 to 45.3] | 25.4 [15.3 to 37.9]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Test type: Other; Risk Difference (RD) = 6.6, 95% CI 2-sided [-9.2 to 22.5] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Progression-free Survival (PFS) Assessed by the Independent Review Committee
Description: Progression-free survival is defined as the time from the date of randomization to the date of first documentation of progressive disease assessed by the Independent Review Committee per RECIST v1.1, or death, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions with an absolute increase of at least 5 mm, or unequivocal progression of existing non-target lesions, or the appearance of any new lesions.
Time Frame: From randomization up to the primary analysis data cutoff date of 01 February 2023; median (range) time on follow-up was 7.4 (0.5 - 20.1) months in Arm A and 6.4 (0.4 - 20.2) months in Arm B.
Population: The Intent-to-Treat (ITT) Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
months | 3.6 [2.7 to 5.1] | 2.8 [1.9 to 6.9]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.64 to 1.59] — Hazard ratio and 95% CIs were estimated using a Cox regression model stratified by the selected stratification factors (ECOG PS score [0 vs 1] and the number of organs with metastases [≤ 1 vs ≥ 2])

5. Secondary Outcome: Progression-free Survival (PFS) Assessed by the Investigator
Description: Progression-free survival is defined as the time from the date of randomization to the date of first documentation of progressive disease assessed by the Investigator per RECIST v1.1, or death, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method.
  Progressive Disease (PD): At least a 20% increase in the size of target lesions with an absolute increase of at least 5 mm, or unequivocal progression of existing non-target lesions, or the appearance of any new lesions.
Time Frame: as for outcome 2
Population: The Intent-to-Treat (ITT) Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
months | 3.4 [1.8 to 5.1] | 3.4 [1.9 to 4.1]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Test type: Other; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.71 to 1.61] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Duration Of Response (DOR) Assessed by the Independent Review Committee
Description: Duration of response is defined as the time from the first determination of an objective response (CR or PR) until the first documentation of progressive disease as assessed by the Independent Review Committee per RECIST v1.1, or death, whichever occurred first.
  Median DOR was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 4
Population: Participants in the Intent-to-Treat Analysis Set who had an objective response per IRC assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 20 | 16
months | 14.6 [7.2 to NA] — Could not be estimated due to the low number of events | NA [4.2 to NA] — Could not be estimated due to the low number of events

7. Secondary Outcome: Duration Of Response (DOR) Assessed by the Investigator
Description: Duration of response is defined as the time from the first determination of an objective response (CR or PR) until the first documentation of progressive disease as assessed by the Investigator per RECIST v1.1, or death, whichever occurred first.
  Median DOR was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 2
Population: Participants in the Intent-to-Treat Analysis Set who had an objective response per Investigator assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 19 | 14
months | 11.3 [5.7 to NA] — Could not be estimated due to the low number of events | NA [4.1 to NA] — Could not be estimated due to the low number of events

8. Secondary Outcome: Disease Control Rate Assessed by the IRC And the Investigator
Description: Disease Control Rate is defined as the percentage of participants who had confirmed CR, PR, or stable disease (SD) assessed by the IRC and the investigator per RECIST v1.1. Response evaluations were performed using computed tomography or MRI approximately every 6 weeks for the first 54 weeks and then every 12 weeks thereafter.
  CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) < 10 mm, and no new lesions.
  PR: At least a 30% decrease in the size of target lesions, with no progression of non-target lesions and no new lesions, or disappearance of target lesions with persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions.
  SD: Neither sufficient shrinkage in size of lesions to qualify for PR nor sufficient increase to qualify for PD, and no new lesions.
  Response (CR or PR) must have been confirmed 4 weeks or later after the first response.
Time Frame: as for outcome 1
Population: The Intent-to-Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
percentage of participants
  Investigator assessment | 61.3 [48.1 to 73.4] | 58.7 [45.6 to 71.0]
  Independent Review Committee | 64.5 [51.3 to 76.3] | 58.7 [45.6 to 71.0]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Disease Control Rate Assessed by the Investigator; Test type: Other; Risk Difference (RD) = 2.7, 95% CI 2-sided [-14.4 to 19.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Disease Control Rate Assessed by the Independent Review Committee; Test type: Other; Risk Difference (RD) = 5.0, 95% CI 2-sided [-11.7 to 21.8] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Clinical Benefit Rate Assessed by the IRC and the Investigator
Description: Clinical benefit rate is defined as the percentage of participants who achieved a confirmed complete response, partial response, or durable stable disease assessed by the IRC and the Investigator per RECIST v1.1. Response evaluations were performed using computed tomography or MRI approximately every 6 weeks for the first 54 weeks and then every 12 weeks thereafter.
  CR: Disappearance of all target and non-target lesions; any pathological lymph nodes (whether target or non-target) < 10 mm, and no new lesions.
  PR: At least a 30% decrease in the size of target lesions, with no progression of non-target lesions and no new lesions, or disappearance of target lesions with persistence of 1 or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits, and no new lesions.
  Durable SD: Stable disease for ≥ 24 weeks. Response (CR or PR) must have been confirmed 4 weeks or later after the first response.
Time Frame: as for outcome 1
Population: The Intent-to-Treat (ITT) Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
percentage of participants
  Investigator Assessment | 33.9 [22.3 to 47.0] | 30.2 [19.2 to 43.0]
  Independent Review Committee | 32.3 [20.9 to 45.3] | 27.0 [16.6 to 39.7]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Clinical Benefit Rate Assessed by the Investigator; Test type: Other; Risk Difference (RD) = 3.9, 95% CI 2-sided [-12.7 to 20.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Clinical Benefit Rate Assessed by the Independent Review Committee; Test type: Other; Risk Difference (RD) = 5.0, 95% CI 2-sided [-11.0 to 21.0] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (GHS)/Quality of Life (QOL) and Physical Functioning Scores
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline, Cycle 5 Day 1 and Cycle 7 Day 1 (each cycle was 3 weeks)
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-C30 at baseline; participants with available data at baseline and the relevant post-baseline visit are included in the analysis at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 50 | 48
score on a scale
  Global Health Status/QOL: Cycle 5: number analyzed (Participants) | 32 | 30
  Global Health Status/QOL: Cycle 5 | 1.7 [-5.6 to 8.9] | -0.1 [-7.5 to 7.4]
  Global Health Status/QOL: Cycle 7: number analyzed (Participants) | 21 | 20
  Global Health Status/QOL: Cycle 7 | 0.3 [-5.6 to 6.1] | -2.8 [-8.8 to 3.2]
  Physical Functioning: Cycle 5: number analyzed (Participants) | 32 | 30
  Physical Functioning: Cycle 5 | -0.5 [-4.3 to 3.3] | 1.2 [-2.8 to 5.2]
  Physical Functioning: Cycle 7: number analyzed (Participants) | 21 | 20
  Physical Functioning: Cycle 7 | -4.4 [-11.2 to 2.5] | -3.9 [-11.0 to 3.3]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Global Health Status/QoL at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; Least Squares (LS) Mean Difference = 1.8, 95% CI 2-sided [-8.4 to 11.9]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Global Health Status/QoL at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = 3.1, 95% CI 2-sided [-5.0 to 11.2]
Statistical Analysis 3: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Physical Functioning at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Superiority; LS Mean Difference = -1.7, 95% CI 2-sided [-7.1 to 3.7]
Statistical Analysis 4: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Physical Functioning at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -0.5, 95% CI 2-sided [-10.3 to 9.3]

11. Secondary Outcome: Change From Baseline in EORTC Quality of Life Oesophageal Cancer Questionnaires 18 (QLQ-OES18) Dysphagia, Eating, Reflux and Pain Scales
Description: The EORTC-QLQ-OES18 is the specific esophageal symptoms module of the QLQ-C30. QLQ-OES18 is comprised of 18 questions grouped into 4 multi-item subscales: Dysphagia (3 items), Eating (4 items), Reflux (2 items), and Pain (3 items) and 6 single item subscales (saliva swallowing, choking, dry mouth, taste, coughing, and talking). Participants indicate the extent to which they have experienced symptoms on a scale from 1 (Not at all) to 4 (Very much). Scores are calculated and transformed to a scale from 0 to 100; higher scores indicate a higher level of symptomatology or problems.
Time Frame: Baseline, Cycle 5 Day 1 and Cycle 7 Day 1 (each cycle was 3 weeks)
Population: Participants in the ITT Analysis Set who completed the EORTC QLQ-OES18 at baseline; participants with available data at baseline and the relevant post-baseline visit are included in the analysis at each time point.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 52 | 48
score on a scale
  Dysphagia: Cycle 5: number analyzed (Participants) | 34 | 30
  Dysphagia: Cycle 5 | -5.9 [-14.2 to 2.4] | 4.1 [-4.7 to 12.8]
  Dysphagia: Cycle 7: number analyzed (Participants) | 22 | 20
  Dysphagia: Cycle 7 | -3.5 [-15.4 to 8.5] | 7.3 [-5.2 to 19.8]
  Eating: Cycle 5: number analyzed (Participants) | 34 | 29
  Eating: Cycle 5 | -1.6 [-6.6 to 3.3] | -1.3 [-6.6 to 4.1]
  Eating: Cycle 7: number analyzed (Participants) | 22 | 20
  Eating: Cycle 7 | -2.8 [-9.1 to 3.6] | 6.6 [-0.2 to 13.4]
  Reflux: Cycle 5: number analyzed (Participants) | 33 | 30
  Reflux: Cycle 5 | 1.9 [-4.6 to 8.3] | -0.4 [-7.1 to 6.4]
  Reflux: Cycle 7: number analyzed (Participants) | 22 | 20
  Reflux: Cycle 7 | 2.7 [-4.8 to 10.1] | 4.0 [-3.8 to 11.8]
  Pain: Cycle 5: number analyzed (Participants) | 33 | 30
  Pain: Cycle 5 | 0.1 [-5.5 to 5.6] | -0.7 [-6.5 to 5.1]
  Pain: Cycle 7: number analyzed (Participants) | 22 | 20
  Pain: Cycle 7 | -2.1 [-7.1 to 3.0] | 3.3 [-2.0 to 8.5]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Dysphagia at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -9.9, 95% CI 2-sided [-21.5 to 1.6]
Statistical Analysis 2: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Dysphagia at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -10.8, 95% CI 2-sided [-27.8 to 6.3]
Statistical Analysis 3: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Eating at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -0.4, 95% CI 2-sided [-7.3 to 6.6]
Statistical Analysis 4: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Eating at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -9.4, 95% CI 2-sided [-18.5 to -0.3]
Statistical Analysis 5: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Reflux at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = 2.3, 95% CI 2-sided [-6.7 to 11.2]
Statistical Analysis 6: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Reflux at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -1.4, 95% CI 2-sided [-11.8 to 9.0]
Statistical Analysis 7: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Pain at Cycle 5. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = 0.7, 95% CI 2-sided [-7.0 to 8.5]
Statistical Analysis 8: Comparison: Arm A: Tislelizumab Plus Ociperlimab vs Arm B: Tislelizumab Plus Placebo; Analysis of Change from Baseline in Pain at Cycle 7. The mixed effect model analysis included the questionnaire score as dependent variable; baseline score, stratification factors, treatment arm, visit, and treatment arm by visit interaction as fixed effects; and visit as a repeated measure, with an unstructured covariance structure; Test type: Other; LS Mean Difference = -5.3, 95% CI 2-sided [-12.3 to 1.7]

12. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study drugs, whether related to study drugs or not.
  An SAE is any untoward medical occurrence that, at any dose:
  * Resulted in death
  * Was life-threatening
  * Required hospitalization or prolongation of existing hospitalization
  * Resulted in disability/incapacity
  * Was a congenital anomaly/birth defect
  * Was considered a significant medical AE by the Investigator based on medical judgement.
  AEs were considered "related" to study drugs if there was evidence to suggest a causal relationship.
  The investigator assessed the severity of each AE reported based upon National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0, where ≥ 3 includes severe or medically significant, life-threatening events or death related to AE.
  Immune-mediated AEs were diagnosed by the investigator.
Time Frame: From first dose of study drug until 30 days after last dose; median duration of treatment was 3.45 months in Tislelizumab + Ociperlimab arm and 2.79 months in the Tislelizumab + Placebo arm.
Population: The Safety Analysis Set included all patients who received ≥ 1 dose of any component of study drugs.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
Number analyzed (Participants) | 62 | 63
Participants
  Any TEAE | 58 | 60
  TEAE ≥ Grade 3 | 28 | 28
  Serious AEs | 27 | 28
  Related SAEs | 13 | 13
  TEAEs Leading to Treatment Discontinuation | 9 | 10
  TEAEs Leading to Death (Excluding Due to Disease Under Study) | 4 | 4
  Any Immune-Mediated AE | 31 | 21
  Immune-Mediated AE ≥ Grade 3 | 8 | 3

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization through the end of study; up to 30 months. AEs are reported from first dose of study drug until 30 days after last dose; median duration of treatment was 3.45 months in Tislelizumab + Ociperlimab arm and 2.79 months in the Tislelizumab + Placebo arm.
Arm/Group | Arm A: Tislelizumab Plus Ociperlimab | Arm B: Tislelizumab Plus Placebo
All-Cause Mortality (participants affected / at risk) | 39/62 | 36/63
Serious Adverse Events (participants affected / at risk) | 27/62 | 28/63
Other Adverse Events (participants affected / at risk) | 57/62 | 54/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab Plus Ociperlimab (N=62) | Arm B: Tislelizumab Plus Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Secondary adrenocortical insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 5 (5)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acquired tracheo-oesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Tislelizumab Plus Ociperlimab (N=62) | Arm B: Tislelizumab Plus Placebo (N=63)
Anaemia (Blood and lymphatic system disorders) | 17 (29) | 20 (25)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 11 (14) | 13 (15)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 3 (5)
Constipation (Gastrointestinal disorders) | 13 (14) | 8 (8)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 4 (5)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (5) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (5)
Oesophageal obstruction (Gastrointestinal disorders) | 3 (3) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 5 (5) | 5 (5)
Asthenia (General disorders) | 5 (6) | 6 (8)
Chest pain (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 8 (8) | 5 (5)
Malaise (General disorders) | 1 (1) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (3) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 4 (6) | 5 (5)
COVID-19 (Infections and infestations) | 6 (7) | 2 (3)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Tuberculosis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 6 (7)
Alanine aminotransferase increased (Investigations) | 4 (7) | 9 (9)
Aspartate aminotransferase increased (Investigations) | 4 (9) | 8 (8)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 2 (3) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 5 (7) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1) | 2 (2)
Blood lactate dehydrogenase increased (Investigations) | 3 (4) | 1 (1)
Blood thyroid stimulating hormone decreased (Investigations) | 0 (0) | 2 (2)
Blood urea increased (Investigations) | 1 (1) | 3 (3)
Electrocardiogram high voltage (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 6 (9) | 3 (3)
Neutrophil count decreased (Investigations) | 2 (5) | 4 (10)
Platelet count decreased (Investigations) | 2 (2) | 3 (3)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 2 (2)
Tri-iodothyronine decreased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 10 (11) | 6 (6)
White blood cell count decreased (Investigations) | 4 (9) | 4 (10)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6) | 11 (12)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyperchloraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (9) | 1 (3)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 9 (14) | 10 (17)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypochloraemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 9 (10) | 7 (8)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (6) | 5 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 13 (17)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 8 (9) | 3 (3)
Hypertension (Vascular disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights

DOCUMENTS (2):
  • Study Protocol (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT04732494/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT04732494/SAP_001.pdf